CLINICAL TRIAL: NCT03957252
Title: Clinical Validation of ClarityDX Prostate as a Reflex Test to Prostate Specific Antigen (PSA) to Refine the Prediction of Clinically-significant Prostate Cancer
Brief Title: Validation of ClarityDX Prostate as a Reflex Test to Refine the Prediction of Clinically-significant Prostate Cancer
Acronym: APCaRI-05
Status: Active, not recruiting | Type: Observational
Sponsor: Nanostics (Industry)
Collaborators: Alberta Prostate Cancer Research Initiative, APCaRI (Unknown); Prostate Cencer Centre, Calgary (Unknown); Alberta Cancer Foundation (Other); Alberta Innovates Health Solutions (Other); Motorcycle Ride for Dad (Unknown); University Hospital Foundation - The Kaye Fund Competition (Unknown); Alberta Precision Laboratories (Unknown); Kipnes Urology Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: APCaRI-05
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: ClarityDX Prostate; Diagnosis; Reflex Test
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Separator Tube (SST) Serum Plasma (EDTA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Cohort: Up to 1400 men from Alberta in addition to up to 2,500 men from external institutions, 40-75 years old, without prior diagnosis of prostate cancer, who have been selected to undergo a prostate biopsy to rule out prostate cancer. Only patients with Total PSA greater than or equal to than 3 ng/mL will be selected to have the ClarityDX Prostate test performed as a reflex test.
  Interventions: Diagnostic Test: Blood test: ClarityDX Prostate
- Validation Cohort: Up to 1400 men from Alberta in addition to up to 2,500 men from external institutions, 40-75 years old, without prior diagnosis of prostate cancer, who have been selected to undergo a prostate biopsy to rule out prostate cancer. Only patients with Tota PSA greater than or equal to 3 ng/mL will be selected to have the ClarityDX Prostate test performed as a reflex test.
  Interventions: Diagnostic Test: Blood test: ClarityDX Prostate

INTERVENTIONS:
Diagnostic Test: Blood test: ClarityDX Prostate — PSA on patients who are suspected to have prostate cancer and will undergo a prostate biopsy. ClarityDX Prostate Risk Score will be compared with biopsy results to assess its predictive accuracy.

SUMMARY:
This study is designed to determine the accuracy of blood test ClarityDX Prostate to predict the results of prostate biopsies in men who have PSA (Prostate Specific Antigen) greater or equal to 3 ng/mL.

DETAILED DESCRIPTION:
The main objective of this study is to validate ClarityDX Prostate as a reflex test to PSA to refine the prediction of clinically-significant prostate cancer in a prospective cohort of men to be recruited in North America when they are scheduled for a biopsy as a result of on an elevated PSA or other suspicion of prostate cancer and in retrospective databases from selected sites in the United States of America and the world.

This prospective training and validation cohort study will consist of up to 2,800 consenting men from Alberta in addition to up to 5,000 men from external institutions, between ages 40-75 (inclusive) years old, without prior diagnosis of prostate cancer, who have been selected to undergo a prostate biopsy to rule out prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males between 40-75 (inclusive) years of age;
2. With and without family history of prostate cancer;
3. No prior prostate cancer diagnosis and who are referred to have a prostate biopsy;
4. Total PSA results >/= 3ng/mL collected within 6m of enrollment;
5. Willing to permit provincial agencies (e.g. Alberta Health Services, Alberta Health, Netcare, Service Alberta or other based on recruitment jurisdiction) to disclose health-related information to study;
6. Undergoing a diagnostic prostate biopsy; and
7. Provided informed consent to participate in the study.

Exclusion Criteria:

1. Unwilling to participate in the study;
2. Unavailable for biopsy procedure in recruitment areas;
3. Not undergoing a prostate biopsy;
4. Prior diagnosis of cancer excluding non-melanoma skin cancer; and/or
5. Under the age of 40 years of age or over the age of 75 years of age.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective training and validation cohort study will consist of up to 2,800 consenting men from Alberta in addition to up to 5,000 men from external institutions, between ages 40-75 (inclusive) years old, without prior diagnosis of prostate cancer, who have been selected to undergo a prostate biopsy to rule out prostate cancer. Only patients with Total PSA >/= 3 ng/mL will be selected to have the ClarityDX Prostate test performed as a reflex test.
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Clinical Performance: prediction of clinically significant prostate cancer at biopsy | 3 years
  Training Phase: Processed clinical features of each patient will be analyzed using machine learning to predict clinically significant prostate cancer, with the output being the ClarityDX Prostate Risk Score.
  Validation Phase: The models created during the Training Phase will be locked down and then used to determine the probability of approximately 1,400 patients in the investigational Validation Phase having clinically significant prostate cancer.
Active Surveillance: prediction of Gleason Grade Group on confirmatory/follow-up biopsies for participants on Active Surveillance | 4 years
MRI: prediction of PI-RADS pre-diagnostic biopsy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Fairey, MD, MSc, Principal Investigator — Kipnes Urology Centre, University of Alberta; Matthew E Hyndman, MD, PhD, Principal Investigator — Southern Alberta Institute of Urology, University of Calgary
Locations (3):
- Johns Hopkins University, Baltimore, Maryland, United States
- Canada (2):
  - Prostate Cancer Centre, Calgary, Alberta
  - Kipnes Urology Centre, Edmonton, Alberta

REFERENCES:
- [Result] Hyndman ME, Paproski RJ, Kinnaird A, Fairey A, Marks L, Pavlovich CP, Fletcher SA, Zachoval R, Adamcova V, Stejskal J, Aprikian A, Wallis CJD, Pink D, Vasquez C, Beatty PH, Lewis JD. Development of an effective predictive screening tool for prostate cancer using the ClarityDX machine learning platform. NPJ Digit Med. 2024 Jun 20;7(1):163. doi: 10.1038/s41746-024-01167-9. PMID 38902526

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03957252/Prot_SAP_001.pdf